CLINICAL TRIAL: NCT01837043
Title: A Randomized Trial of Early Conversion From Calcineurin Inhibitors (CNI) to Belatacept in Renal Transplant Recipients With Delayed and Slow Graft Function
Brief Title: Early Conversion From CNI to Belatacept in Renal Transplant Recipients With Delayed and Slow Graft Function
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nair, Vinay, D.O. (Individual)
Collaborators: Icahn School of Medicine at Mount Sinai (Other); Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IM103-057; 13-00174 (Other: Mount Sinai PPHS)
Record Dates: First submitted 2013-04-16; First posted 2013-04-22 (Estimated); Last update posted 2017-01-30 (Estimated); Status verified 2017-01

CONDITIONS: Delayed Graft Function; Kidney Transplant
Keywords: Delayed Graft Function; Renal Transplantation; Kidney Transplant
MeSH Terms: conditions — Delayed Graft Function | interventions — Abatacept; Calcineurin Inhibitors; Tacrolimus; Cyclosporine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Belatacept (Experimental): Subjects will be converted from standard of care CNI therapy to Belatacept 10 mg/kg IV on post renal transplant Day 7 (+/- 3 days). As suggested in the package insert for de novo dosing, further dosing of belatacept will be given as 10 mg/kg IV at weeks 2, 4, 8 and 12 then 5 mg/kg at week 16 and then every 4 weeks (+/- 5 days) through week 52. CNI will be stopped during the first belatacept infusion.
  Interventions: Drug: Belatacept
- Calcineurin Inhibitor (Active Comparator): Patients randomized to this arm will remain on the current CNI as prescribed by post-transplant standard of care therapy.
  Interventions: Drug: Calcineurin Inhibitor

INTERVENTIONS:
Drug: Belatacept
  Other Names: Nulojix
  Arms: Belatacept
Drug: Calcineurin Inhibitor
  Other Names: Prograf, Tacrolimus, Cyclosporine
  Arms: Calcineurin Inhibitor

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of conversion from a calcineurin inhibitor (tacrolimus or cyclosporine) immunosuppression therapy to Nulojix® (belatacept) immunosuppression therapy in patients with delayed (DGF) or slow graft function (SGF) following kidney transplantation. Patients at risk for SGF or DGF will be consented at the time of kidney transplantation. On post-op Day 5 the patient will be assessed, if they have developed SGF or DGF they will be randomized to convert to Belatacept or continue on their CNI regimen. Up to 20 subjects who do not develop DGF will be followed as control subjects. Seventy randomized subjects will be followed for a total of 14 months with a renal biopsy at Month 12 post transplant.

Research Hypotheses:

Primary Hypotheses:

* Kidneys with slow or delayed graft function are more susceptible to acute and long-term CNI toxicity
* Kidneys converted from calcineurin inhibitor based therapy to belatacept will achieve a more rapid recovery from post-ischemic acute tubular necrosis (ATN) and will have improved 1 year calculated GFR.

Key Secondary Hypotheses:

* Renal Histology: Belatacept converted patients will have a lower chronic allograft damage index (CADI) score and lower interstitial fibrosis and tubular atrophy (IF/TA) score as calculated by Banff criteria at 1 year post- transplant
* Biomarker Analysis: Biomarker analysis (clusterin) measured in serial urine collections can 1) directly assess CNI induced kidney injury and 2) improve the prediction of patients that benefit in early belatacept conversion.

ELIGIBILITY:
Inclusion Criteria:

* Before any study procedures are performed, subjects will have the details of the study described to them, and they will be given a written informed consent document to read. Then, if subjects consent to participate in the study, they will indicate that consent by signing and dating the informed consent document in the presence of study personnel.
* All patients (> 18 years) who have received a deceased donor transplant and are at risk for SGF/DGF will be studied
* All gender and ethnicities will be considered in this study
* At risk for SGF/DGF is defined as:

  * ECD (Extended Criteria Donor) donor kidney recipients
  * ECD is defined as a donor over the age of 60 or age 50 to 60 with 2 of the following risk factors:
* Terminal creatinine > 1.5 mg/dL
* History of Hypertension
* Death due to cerebrovascular accident

  * Donations after cardiac death (DCD) kidney recipients
  * Donor organs with an actual cold ischemia time (CIT) > 19 hours
  * Recipients of donor organs with a terminal creatinine > 1.5 mg/dL
* Only patients who receive Thymoglobulin induction and CNI maintenance at time of randomization will be considered for the study
* Men and women, 18 to 70 years of age
* Reproductive status: Definition of Women of Child-Bearing Potential (WOCBP). WOCBP comprises women who have experienced menarche and who have not undergone successful surgical sterilization (hysterectomy, bilateral tubal ligation, or bilateral oophorectomy) or who are not post-menopausal.

Post-menopause is defined as:

* Women who have had amenorrhea for >= 12 consecutive months (without another cause) and who have a documented serum follicle-stimulating hormone (FSH)level > 35 mIU/mL
* Women who have irregular menstrual periods and a documented serum FSH level > 35 mIU/mL
* Women who are taking hormone replacement therapy

The following are WOCBP:

* Women using the following methods to prevent pregnancy: oral contraceptives, other hormonal contraceptives (vaginal products, skin patches, or implanted or injectable products), or mechanical products such as intrauterine devices or barrier methods (diaphragm, condoms, spermicides).
* Women who are practicing abstinence
* Women who have a partner who is sterile (due to vasectomy)
* WOCBP must be using an acceptable method of contraception to avoid pregnancy throughout the study and for up to 8 weeks after the last dose of study drug in such a manner that the risk of pregnancy is minimized
* WOCBP must have a negative serum or urine pregnancy test result (minimum sensitivity 25 IU/L or equivalent units of HCG) within 24 hours before the first dose of study drug.
* Women must not be breast-feeding
* Sexually active fertile men must use effective birth control if their partners are WOCBP

Exclusion Criteria:

* Seronegative or unknown EBV (Epstein Barr Virus) serostatus (due to the risk of posttransplant lymphoproliferative disorder, PTLD) predominantly involving the central nervous system
* Patients with tuberculosis who have not been treated for latent infection
* Patients at high risk for polyoma virus-associated nephropathy, which is mostly due to BK virus infection
* Rejection episode before randomization
* Anatomic cause of SGF/DGF such as urinary leak, obstruction or thrombosis
* Patients with a prior or concurrent non-renal solid organ transplant
* Patients with living donor kidneys
* Patients with pediatric kidneys (age of less than 5 years)
* Dual kidney transplants (from the same donor)
* Immunologically high risk patients with a positive crossmatch pre- transplantation or donor specific antibody (DSA) > 5000 MFI
* ABO Incompatible transplantation
* Patients with HIV
* Subjects with any active infection or other contraindication that would normally exclude transplantation
* Patients with a history of malignancy in the last 5 years except non- melanoma skin cancer
* Baseline white blood cell count less than 2,000
* Baseline hemoglobin less than 8 g/dL
* Patients with prior allergic reactions to belatacept
* Patients with prior allergic reactions to thymoglobulin
* Sex and Reproductive status - see WOCBP information in inclusion above
* Subjects currently receiving immunosuppressive agent(s) for other indications such as an autoimmune disease or subjects with comorbidities that treatment with such agents are likely during the trial.
* Subjects who have used any investigational drug within 30 days prior to the Day 1 visit
* Subjects previously treated with belatacept
* Prisoners or subjects who are involuntarily incarcerated
* Subjects who are compulsorily detained for treatment of either a psychiatric or physical (e.g. infectious disease) illness.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2013-06; Primary Completion 2017-06 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
cGFR | 12 months
  Serum creatinine will be checked at each study visit from which GFR will be calculated. 12 month 4 variable MDRD calculated GFR will be compared between the belatacept conversion group and the calcineurin inhibitor group.

SECONDARY OUTCOMES:
Renal Histology | 12 months
  Chronic Allograft Damage Index (CADI) and Interstitial Fibrosis/Tubular Atrophy (IFTA) renal pathology scores will be assessed by a local pathologist. CADI and IF/TA will be recorded at baseline (reperfusion biopsy) and at the 1 year protocol biopsy. The average progression of CADI and IF/TA will be compared in both groups and the average absolute CADI and IF/TA scores will be compared in both groups at 1 year post transplant.
Biomarker profile | 12 months
  The results of urine biomarkers (clusterin) will be correlated with the development of the primary and secondary endpoints in both groups. In this manner the investigators will be able to understand which genes/proteins are primarily altered by injury and assess how belatacept affects this process.
Duration of Delayed (or slow) Graft Function | 12 months
  The average duration of DGF/SGF will be compared in both belatacept and CNI groups
Incidence of Acute Rejection | 12 months
  Acute rejection by month 12 will be assessed by a local pathologist using the Banff 97 working classification of kidney transplant pathology. All biopsies will be interpreted locally for purposes of the study.
New Onset Diabetes | 12 months
  Subjects will be evaluated for post-transplant diabetes at visits after week 4.
Blood Pressure Control | 12 months
  Subjects are to be evaluated at each clinic visit to assess the need for adjustment of antihypertensive medication in order to achieve a BP of < 130/80 mmHg. Average systolic and diastolic blood pressure in both groups at Month 12, number of antihypertensive medications and change in intensity of hypertension treatment will be observed.
Dyslipidemia | 12 months
  Cholesterol levels in both groups, number of patients on dyslipidemic therapy at month 12 and change in intensity of dyslipidemia therapy will be observed
Graft Survival | 12 Months
  Graft survival will be observed in both groups and compared at 12 months post-transplant
Patient survival | 12 months
  Patient survival will be observed in both groups and compared at 12 months post-transplant

CONTACTS AND LOCATIONS:
Overall Officials: Vinay Nair, D.O., Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Mount Sinai School of Medicine Recanati/Miller Transplantation Institute, New York, New York, United States